CLINICAL TRIAL: NCT02565771
Title: Evaluation of the Improvement of Autonomic Nervous System by a Physical Rehabilitation Program Adapted to Adulthood After Chemotherapy or Radiotherapy in Childhood
Acronym: SALTO_GyV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1208137; 2012-A01220-43 (Other: ANSM)
Record Dates: First submitted 2015-09-30; First posted 2015-10-01 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Cancer; Sequels; Complications
Keywords: Childhood cancer; Cancer; Sequels; Surgery; Complications; Chemotherapy; Radiotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young adult survivors of childhood cancer: Adults treated for childhood cancer in Rhône-Alpes region in France between 1987 and 1992 with deregulation ANS or autonomic imbalance.
  Interventions: Other: Adapted physical activity

INTERVENTIONS:
Other: Adapted physical activity — The adapted physical activity is done by Education Physique et Gymnastique Volontaire (EPGV) centres.

SUMMARY:
Survival rate of childhood cancers is now reaching 80%. However, early or late complications related to surgery, chemotherapy and radiotherapy remain high and greatly increase the risk of late mortality.

Health of individuals is closely correlated to the stability of the autonomic nervous system (ANS), a key system for maintaining homeostasis in any living species. Efficient computer tools allowed the opportunity to assess the intrinsic autonomic regulation of the ANS either directly or at a later time by an analysis of the heart rate variability (HRV). These tools have become very powerful predictors of cardiovascular morbidity and neurological aging. Physical endurance training improves both maximal aerobic capacity and ANS activity.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate improvement of ANS parameters after 6 months of adapted physical activity in adults treated for childhood cancer in Rhône-alpes region in France who have deregulation ANS or autonomic imbalance.

ELIGIBILITY:
Inclusion Criteria:

* Included in the SALTO_SNA study (NCT01574196)
* Alteration of the autonomic nervous system activity or deregulation of the sympatho-vagal balance

Exclusion Criteria:

* Written consent form
* Left ventricular dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults treated for childhood cancer in Rhône-Alpes region in France between 1987 and 1992 with deregulation ANS or autonomic imbalance.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Autonomic nervous system activity | At 6 months
  The autonomic nervous system activity is classified in sympatho-vagal equilibrium as "normal", "altered" or "severely abnormal".
  For this classification, we need the values obtained for some temporal indices (Standard Deviation NN intervals (SDNN), Root Mean Square of Successive Differences (RMSSD)) and frequencies (Ptot, High Frequency (HF), Low Frequency (LF) , Very-Low Frequency (VLF), ratio LF / HF) compared to validated standards for the age (mean +/- standard deviation).

SECONDARY OUTCOMES:
Daily activity questionnaire | At 6 months
Quality of Life Questionnaire | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Claire BERGER, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No